CLINICAL TRIAL: NCT00963872
Title: MT2008-15: Transplantation of Unrelated Donor Umbilical Cord Blood in Patients With Hematological Malignancies Using a Nonmyeloablative Preparative Regimen and Priming With Complement 3a Fragment (C3a)
Brief Title: Donor Umbilical Cord Blood Transplant After Fludarabine Phosphate, Cyclophosphamide, and Total-Body Irradiation in Treating Patients With High-Risk Hematologic Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy after interim analysis
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008UC097; MT2008-15 (Other: Blood and Marrow Transplantation Program); 0809M46361 (Other: IRB, University of Minnesota); RC1HL099447 (NIH)
Record Dates: First submitted 2009-08-21; First posted 2009-08-24 (Estimated); Results first posted 2015-11-10 (Estimated); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Leukemia; Lymphoma; Multiple Myeloma; Myelodysplastic Syndromes
MeSH Terms: conditions — Leukemia; Lymphoma; Multiple Myeloma; Myelodysplastic Syndromes | interventions — Cyclophosphamide; fludarabine phosphate; Whole-Body Irradiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Complement Fragment 3A - Small Cell Dose (Experimental): Patients who received complement fragment 3a (C3a) priming of the UCB unit with the smaller cell dose following preparation regimen and radiation.
  Interventions: Drug: cyclophosphamide; Drug: fludarabine phosphate; Radiation: Total body irradiation; Biological: Umbilical cord blood unit with C3a fragment; Biological: Unmanipulated UCB Unit
- Complement Fragment A - Larger Cell Dose (Experimental): Patients who received complement fragment 3a (C3a) priming of the UCB unit with the larger cell dose.
  Interventions: Drug: cyclophosphamide; Drug: fludarabine phosphate; Radiation: Total body irradiation; Biological: Umbilical cord blood unit with C3a fragment; Biological: Unmanipulated UCB Unit

INTERVENTIONS:
Drug: cyclophosphamide — 50 mg/kg intravenously (IV) over 2 hours on Day -6.
  Other Names: Cytoxan
Drug: fludarabine phosphate — 40 mg/m^2 over 1 hour on Days -6 through -2.
  Other Names: Fludara
Radiation: Total body irradiation — 200 cGy on Day -1
Biological: Umbilical cord blood unit with C3a fragment — On Day 0, the C3a primed UCB unit will be infused intravenously SECOND, within 30 minutes of the completion of the infusion of the unmanipulated UCB unit, through a central line without in-line filtration in a manner identical to the unmanipulated UCB unit.
Biological: Unmanipulated UCB Unit — On Day 0, the unmanipulated UCB unit will be infused FIRST through a central line without in-line filtration per institutional guidelines.

SUMMARY:
RATIONALE: Giving low doses of chemotherapy and total-body irradiation before a donor umbilical cord blood transplant helps stop the growth of cancer cells. It may also stop the patient's immune system from rejecting the donor's stem cells. The donated stem cells may replace the patient's immune cells and help destroy any remaining cancer cells (graft-versus-tumor effect).

PURPOSE: This phase I trial is studying the safety of donor umbilical cord blood transplant after fludarabine phosphate, cyclophosphamide, and total-body irradiation in treating patients with high-risk hematologic cancer (now closed).

The Phase II part of this trial is studying whether priming one of two UCB units with C3a facilitates engraftment of the treated unit.

DETAILED DESCRIPTION:
OUTLINE:

* Nonmyeloablative preparative regimen: Patients receive fludarabine phosphate IV over 1 hour on days -6 to -2 and cyclophosphamide IV over 2 hours on day -6. Patients then undergo total-body irradiation on day -1. Some patients also receive anti-thymocyte globulin IV every 12 hours on days -6, -5, and -4.
* Umbilical cord blood (UCB) transplantation: Patients undergo unmanipulated UCB transplantation followed by complement 3a fragment primed UCB transplantation on day 0.

Treatment for graft-vs-host disease prophylaxis is also given.

After completion of study therapy, patients are followed up periodically for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Disease Criteria

  * Acute Leukemias: Must be in remission by morphology (<5% blasts). Note cytogenetic relapse or persistent disease without morphologic relapse is acceptable. Also a small percentage of blasts that is equivocal between marrow regeneration vs. early relapse are acceptable provided there are no associated cytogenetic markers consistent with relapse. (See exclusion criteria for more detailed definition)
  * Acute myeloid leukemia: high risk CR1 (as evidenced by preceding myelodysplastic syndrome (MDS), high risk cytogenetics such as those associated with MDS or complex karyotype, > 2 cycles to obtain complete remission (CR) or erythroblastic and megakaryocytic); second or greater CR.
  * Acute lymphoblastic leukemia/lymphoma: high risk CR1 as evidenced by high risk cytogenetics (e.g. t(9;22, t(1;19), t(4;11), other MLL rearrangements) or > 1 cycle to obtain CR; second or greater CR.
  * Burkitt's lymphoma in CR2 or subsequent CR
  * Natural Killer cell malignancies
  * Myeloproliferative syndromes/diseases: Chronic myelogenous leukemia (CML) in chronic or accelerated phase but patients must have failed or been intolerant to Imatinib mesylate. EXCLUDED: CML in refractory blast crisis, myelofibrosis, polycythemia vera, and essential thrombocytosis.
  * Myelodysplastic Syndrome: any subtype including refractory anemia (RA) if severe pancytopenia, high risk complex cytogenetics or International Prognostic Scoring System (IPSS) ≥ intermediate-2 (Int-2). Blasts must be less than 5%. If 5% or more requires therapy pre-transplant to reduce blast count to ≤5%. Patients who receive single agent 5-azacytidine, decitabine or immunomodulating drugs are eligible.
  * Large-cell lymphoma, Hodgkin's lymphoma and multiple myeloma: patients with chemotherapy sensitive disease that has failed or who are ineligible for an autologous transplant. Patients are eligible for umbilical cord blood (UCB) transplantation if there is no evidence of progressive disease by imaging modalities and/or biopsy. Persistent PET activity, though possibly related to lymphoma, IS NOT an exclusion criterion in the absence of computated tomography (CT) changes in size indicating progression. Large-cell and Hodgkin's lymphoma that is progressive on salvage therapy is NOT eligible. Patients with stable disease are eligible for transplantation if the largest residual nodal mass is < 5 cm (approximately). For patients who have responded to preceding therapy, the largest residual mass must represent a 50% reduction and be < 7.5 cm (approximately).
  * Chronic lymphocytic leukemia/small lymphocytic lymphoma (CLL/SLL), marginal zone B-cell lymphoma, follicular lymphoma which have progressed after at least two prior therapies. Patients with bulky disease should be considered for debulking chemotherapy before transplant. Patients with refractory disease are eligible, unless has bulky disease and an estimated tumor doubling time of less than one month. Patients with stable disease are eligible for transplantation if the largest residual nodal mass is < 5 cm (approximately). For patients who have responded to preceding therapy, the largest residual mass must represent a 50% reduction and be < 7.5 cm (approximately).
  * Lymphoplasmacytic lymphoma, mantle-cell lymphoma, prolymphocytic leukemia are eligible after initial therapy if chemotherapy sensitive. Mantle-cell lymphoma that is progressive on salvage therapy is NOT eligible. Patients with stable disease are eligible for transplantation if the largest residual nodal mass is < 5 cm (approximately). For patients who have responded to preceding therapy, the largest residual mass must represent a 50% reduction and be < 7.5 cm (approximately).
* Umbilical Cord Blood Graft Selection - Two UCB units will be compose the graft, and each unit must be a 4-6 HLA-A, B, DRB1 antigen match to each other, as well as a 4-6 antigen match to the recipient. The combined cryopreserved nucleated cell dose of the 2 units must be ≥ 3 X 10^7/kg with each unit having a minimum cell dose of 1.5 X 10^7/kg. UCB units will be selected according to a common umbilical cord blood graft selection algorithm
* Performance Status - adequate performance status defined as Karnofsky score ≥ 60
* Age 18 to 70 years of age; patients ≥ 70 but ≤ 75 years are eligible if the co-morbidity score is ≤ 2
* Organ Function

  * Cardiac: Left ventricular ejection fraction > 35%; absence of decompensated congestive heart failure; absence of uncontrolled arrhythmia
  * Pulmonary: DLCO > 30% of predicted; absence of O2 requirements
  * Hepatic: ALT, AST, alkaline phosphatase and bilirubin < 5 x upper limit of normal
  * Renal: Creatinine ≤ 2 mg/dl (patients with a creatinine > 1.2 or history of renal dysfunction must have calculated glomerular filtration rate (GFR) > 40 mL/min/1.73m2)
  * If recent mold infection e.g. Aspergillus - must have minimum of 30 days of appropriate treatment before transplant and infection controlled and be cleared by Infectious Disease.
  * The following conditions must be met:

    * If prior myeloablative autologous transplant, must be > 3 months but ≤ 12 months from transplant OR have received at least 2 cycles of multi-agent or highly immunosuppressive chemotherapy (i.e. induction for acute leukemia) within the 3 months preceding this study. OR
    * If neither prior myeloablative autologous transplant ≤ 12 months from transplant nor have received at least 2 cycles of multi-agent or highly immunosuppressive chemotherapy (i.e. induction for acute leukemia) within the 3 months preceding this study, patients are eligible as long as they receive equine anti-thymocyte globulin as part of the conditioning regimen.

Exclusion Criteria:

* Patients who have an available, medically suitable, 5-6/6 HLA-A, B, DRB1 matched sibling donor
* Patients who are eligible for autologous transplantation
* Prior allogeneic transplant
* Acquired or inherited bone marrow failure syndromes such as aplastic anemia and Fanconi anemia
* Pregnant or breast feeding
* Evidence of HIV infection or known HIV positive serology
* Current uncontrolled serious infection
* Active central nervous system malignancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2010-03; Primary Completion 2012-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claudio G. Brunstein, MD, PhD, Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- University of Minnesota Medical Center - Fairview, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited at the time of clinic visit or hospitalization. Patients that were considered for umbilical cord transplant were approached with the study.
Pre-assignment Details: Subjects that were eligible for umbilical cord transplant were considered for the study.
Period: Overall Study
Arm/Group | Complement Fragment 3A - Small Cell Dose | Complement Fragment A - Larger Cell Dose
Started | 25 | 6
Completed | 24 | 5
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Population: Two patients were unevaluable because 1 bag broke so only 1 cord was available. One subject never received the C3a.
Groups:
- Total: Total of all reporting groups
Arm/Group | Complement Fragment 3A - Small Cell Dose | Complement Fragment A - Larger Cell Dose | Total
Number analyzed (Participants) | 25 | 6 | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 5 | 24
  >=65 years | 6 | 1 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 55 (13.0) | 50 (15.7) | 54 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 2 | 11
  Male | 16 | 4 | 20
Region of Enrollment [Number; unit: participants]
  United States | 25 | 6 | 31

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With the Complement 3a (C3a) Unit Predominating
Description: Efficacy of the pre-incubation of one of two umbilical cord blood (UCB) units with C3a as part of a unrelated donor double UCB nonmyeloablative transplantation in patients with high-risk hematological malignancies.
Time Frame: Day 180
Population: Two patients were unevaluable - one, because 1 bag of cord blood broke leaving only 1 cord available, and one subject never received the C3a.
Measure: Number; unit: participants
Arm/Group | Complement Fragment 3A - Small Cell Dose | Complement Fragment A - Larger Cell Dose
Number analyzed (Participants) | 24 | 5
participants | 9 | 5

2. Secondary Outcome: Neutrophil Engraftment
Description: Achieving 500 neutrophils/uL by day 42.
Time Frame: Day 42
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Complement Fragment 3A - Small Cell Dose | Complement Fragment A - Larger Cell Dose
Number analyzed (Participants) | 24 | 5
participants | 22 | 5

3. Secondary Outcome: Donor Chimerism in Blood
Description: Percentage of donor DNA present in the peripheral blood
Time Frame: Day 28
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of donor DNA
Arm/Group | Complement Fragment 3A - Small Cell Dose | Complement Fragment A - Larger Cell Dose
Number analyzed (Participants) | 24 | 5
percentage of donor DNA | 92 (15) | 96 (8)

4. Secondary Outcome: Incidence of Grades II-IV Graft-vs-host Disease
Description: Development of graft-versus-host disease through day 100.
Time Frame: Day 0 through Day 100
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Complement Fragment 3A - Small Cell Dose | Complement Fragment A - Larger Cell Dose
Number analyzed (Participants) | 24 | 5
participants | 8 | 1

5. Secondary Outcome: Non-Relapse Mortality
Description: Deaths not due to relapse.
Time Frame: Day 180
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Complement Fragment 3A - Small Cell Dose | Complement Fragment A - Larger Cell Dose
Number analyzed (Participants) | 24 | 5
participants | 3 | 0

6. Secondary Outcome: Overall Survival
Description: Survival (alive) from transplantation to last follow-up.
Time Frame: Day 360
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Complement Fragment 3A - Small Cell Dose | Complement Fragment A - Larger Cell Dose
Number analyzed (Participants) | 24 | 5
participants | 14 | 5

7. Secondary Outcome: Bone Marrow Chimerism
Description: Percentage of donor DNA in the bone marrow.
Time Frame: Day 21
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of donor DNA
Arm/Group | Complement Fragment 3A - Small Cell Dose | Complement Fragment A - Larger Cell Dose
Number analyzed (Participants) | 24 | 5
percentage of donor DNA | 84 (25) | 89 (23)

8. Secondary Outcome: Chronic Graft-Versus-Host Disease
Description: Patients who developed chronic graft-versus-host disease.
Time Frame: Day 360
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Complement Fragment 3A - Small Cell Dose | Complement Fragment A - Larger Cell Dose
Number analyzed (Participants) | 24 | 5
participants | 0 | 0

9. Secondary Outcome: Relapse of Disease
Description: Patients who developed disease relapse after transplantation.
Time Frame: Day 360
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Complement Fragment 3A - Small Cell Dose | Complement Fragment A - Larger Cell Dose
Number analyzed (Participants) | 24 | 5
participants | 10 | 0

10. Secondary Outcome: Disease Progression
Description: Patients who developed disease progression after transplantation.
Time Frame: Day 360
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Complement Fragment 3A - Small Cell Dose | Complement Fragment A - Larger Cell Dose
Number analyzed (Participants) | 24 | 5
participants | 0 | 0

11. Secondary Outcome: Platelet Recovery
Description: Number of patients with >20,000 platelets/uL by day 180
Time Frame: Day 180
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Complement Fragment 3A - Small Cell Dose | Complement Fragment A - Larger Cell Dose
Number analyzed (Participants) | 24 | 5
participants | 19 | 5

12. Secondary Outcome: Donor Chimerism in Blood
Description: Percentage of donor DNA present in the peripheral blood
Time Frame: Day 60
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of donor DNA
Arm/Group | Complement Fragment 3A - Small Cell Dose | Complement Fragment A - Larger Cell Dose
Number analyzed (Participants) | 24 | 5
percentage of donor DNA | 91 (23) | 97 (4)

13. Secondary Outcome: Incidence of Grades III-IV Graft-vs-host Disease
Description: Development of graft-versus-host disease by day 100.
Time Frame: 0 to 100 days
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Complement Fragment 3A - Small Cell Dose | Complement Fragment A - Larger Cell Dose
Number analyzed (Participants) | 24 | 5
participants | 2 | 0

14. Secondary Outcome: Non-relapse Mortality
Description: Deaths not due to relapse.
Time Frame: Day 360
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Complement Fragment 3A - Small Cell Dose | Complement Fragment A - Larger Cell Dose
Number analyzed (Participants) | 24 | 5
participants | 3 | 0

15. Secondary Outcome: Overall Survival at Day 720
Description: Survival (alive) from transplantation to last follow-up at day 720.
Time Frame: 720 days
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Complement Fragment 3A - Small Cell Dose | Complement Fragment A - Larger Cell Dose
Number analyzed (Participants) | 24 | 5
participants | 13 | 5

16. Secondary Outcome: Relapse of Disease
Description: Patients who developed disease relapse after transplantation.
Time Frame: Day 720
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Complement Fragment 3A - Small Cell Dose | Complement Fragment A - Larger Cell Dose
Number analyzed (Participants) | 24 | 5
participants | 11 | 1

17. Secondary Outcome: Disease Progression
Description: Patients who developed disease progression after transplantation.
Time Frame: Day 720
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Complement Fragment 3A - Small Cell Dose | Complement Fragment A - Larger Cell Dose
Number analyzed (Participants) | 24 | 5
participants | 0 | 0

18. Secondary Outcome: Donor Chimerism
Description: Percentage of donor DNA in the bone marrow.
Time Frame: Day 100
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of donor DNA
Arm/Group | Complement Fragment 3A - Small Cell Dose | Complement Fragment A - Larger Cell Dose
Number analyzed (Participants) | 24 | 5
percentage of donor DNA | 90 (22) | 94 (19)

19. Secondary Outcome: Donor Chimerism
Description: Percentage of donor DNA in the bone marrow.
Time Frame: Day 180
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of donor DNA
Arm/Group | Complement Fragment 3A - Small Cell Dose | Complement Fragment A - Larger Cell Dose
Number analyzed (Participants) | 24 | 5
percentage of donor DNA | 99 (3) | 100 (0)

20. Secondary Outcome: Donor Chimerism
Description: Percentage of donor DNA in the bone marrow.
Time Frame: Day 360
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of donor DNA
Arm/Group | Complement Fragment 3A - Small Cell Dose | Complement Fragment A - Larger Cell Dose
Number analyzed (Participants) | 24 | 5
percentage of donor DNA | 93 (19) | 100 (0)

ADVERSE EVENTS:
Time Frame: 100 days after umbilical cord blood transplant
Arm/Group | Complement Fragment 3A - Small Cell Dose | Complement Fragment A - Larger Cell Dose
Serious Adverse Events (participants affected / at risk) | 21/24 | 5/5
Other Adverse Events (participants affected / at risk) | 24/24 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Complement Fragment 3A - Small Cell Dose (N=24) | Complement Fragment A - Larger Cell Dose (N=5)
Blood and lymphatic disorders- Other (Blood and lymphatic system disorders) | 10 (10) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Death NOS (General disorders) | 2 (2) | 0 (0) — Death due to disease
Fever (General disorders) | 5 (5) | 0 (0)
Infusion related reaction (General disorders) | 0 (0) | 1 (1)
Catheter related infection (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 2 (2) | 0 (0)
Confusion (Psychiatric disorders) | 2 (2) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal and urinary disorders- Other (Renal and urinary disorders) | 1 (1) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleuritic plan (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Complement Fragment 3A - Small Cell Dose (N=24) | Complement Fragment A - Larger Cell Dose (N=5)
Rash (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Hypertension (Blood and lymphatic system disorders) | 24 (24) | 4 (4)
Sinus tachycardia (Cardiac disorders) | 2 (2) | 1 (1)
Neurologic disorder (Nervous system disorders) | 4 (4) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 7 (7) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes